CLINICAL TRIAL: NCT01685528
Title: VA Home-Based Emotional Learning With Practical Skills (VA-HELPS): Treatment for Depressed and/or Anxious Rural Veterans in Home-Based Primary Care
Brief Title: VA Home-Based Emotional Learning With Practical Skills
Acronym: VA-HELPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melinda Stanley, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30655
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Geriatric; Veteran
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT (Experimental)
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — 6-8 weekly sessions of CBT, 1 of which is in person with the rest being over the telephone
  Other Names: Cognitive Behavior Treatment, Cognitive Behavior Therapy

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of providing evidence-based, person-centered, culturally tailored treatment for anxiety and/or depression via telephone to rural Veterans receiving home-based primary care.

DETAILED DESCRIPTION:
VA-HELPS will include flexibility in both content and delivery to meet the needs of Home Based Primary Care (HBPC) Veterans. Content will be modular to meet the needs of both anxious and depressed participants. Modular skills-based treatment has been used successfully with a range of clinical problems (Chorpita et al., 2004; Henin et al., 2001; Wetherell et al., 2009, 2011), including our own group's work treating generalized anxiety disorder (GAD) in primary care (Calleo et al., in press) and anxiety-depression in patients with chronic illness (Cully et al., 2010). To further support a patient-centered treatment approach, patients will have the opportunity to include R/S. Research points to the importance of R/S in coping with illness, with 50-90% of patients reporting using their belief systems to enhance coping skills (Koenig & Adams, 2008). Along with content modifications, delivery of treatment should complement the needs of HBPC Veterans. Providing one initial in-home session, followed by telephone contact for subsequent sessions, allows cost effectiveness to be taken into consideration; and greater numbers of rural HBPC patients will have access to the intervention.

Treatment will involve approximately 6 to 8 weekly sessions lasting approximately 30-40 minutes each. After the first in-person session, all sessions will be delivered via telephone. At least one booster call (15-20 minutes) will occur during the month following completion of active treatment. All participants will complete assessments at baseline, 8 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Part of Home-Based Primary Care
* Reside in a rural community, as defined by the US Census Bureau
* Symptoms of anxiety and/or depression

Exclusion Criteria:

* Significant cognitive impairment
* Active suicidal intent
* Current uncontrolled psychosis, bipolar, or substance-abuse disorders within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Geriatric Anxiety Inventory | 12 weeks
Penn State Worry Questionnaire (PSWQ-A) | 12 weeks
Generalized Anxiety Disorder-7 | 12 weeks

SECONDARY OUTCOMES:
SF-12 Health Survey | 12 weeks
Brief RCOPE | 12 weeks
  A measure of positive and negative forms of religious coping
Client Satisfaction Questionnaire | 12 weeks
Patient Health Questionnaire-9 | 12 weeks
Geriatric Depression Scale | 12 weeks
Working Alliance Inventory | 12 weeks
Brief Multidimensional Measure of Religiousness and Spirituality | 12 weeks
Insomnia Severity Index | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A Stanley, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Center for Quality of Care and Utilization Studies, Houston, Texas, United States